CLINICAL TRIAL: NCT00000784
Title: A Study of Psychosocial and Behavioral Determinants of Differential Rates of Participant Compliance in CPCRA Protocols
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPCRA 012; 11564 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- A: Consenting patients newly enrolled in either CPCRA 007 or CPCRA 006

SUMMARY:
To examine, in patients enrolled in protocols CPCRA 006 and/or 007, the relationship between patient compliance and demographic, psychosocial, and lifestyle characteristics and Health Belief Model premises (i.e., patient's perception of susceptibility to and severity of disease and perception of benefits and barriers to a particular treatment) in order to design more effective intervention protocols.

Patient noncompliance can influence the statistical findings of a clinical study, possibly resulting in an incorrect assessment of the effects of the investigational therapeutic agent. Since the special populations targeted by the CPCRA for inclusion in HIV-related clinical research do not typify those traditionally included in clinical trials or compliance research, it is necessary to elucidate and examine the special needs of these populations and to determine the extent to which these needs manifest themselves as potential barriers to protocol compliance.

DETAILED DESCRIPTION:
Patient noncompliance can influence the statistical findings of a clinical study, possibly resulting in an incorrect assessment of the effects of the investigational therapeutic agent. Since the special populations targeted by the CPCRA for inclusion in HIV-related clinical research do not typify those traditionally included in clinical trials or compliance research, it is necessary to elucidate and examine the special needs of these populations and to determine the extent to which these needs manifest themselves as potential barriers to protocol compliance.

Patients who are enrolled on protocols CPCRA 006 and/or 007 are given a baseline questionnaire to complete during the enrollment visit for the qualifying treatment protocol. The survey concerns the patient's work, primary language, support systems, residence status, perception of disease and treatments, and substance use. At 4-month follow-up visits, patients are asked to complete a self-report questionnaire, which assesses the patient's perceptions of difficulties in protocol compliance requirements, clinic/office visits, and health beliefs. The duration of patients on this study will be defined by the qualifying protocol requirements.

ELIGIBILITY:
Patients must meet the following criteria:

* New enrollment on CPCRA 006 or CPCRA 007.
* Life expectancy of at least 6 months.
* Willing and able, in clinician's opinion, to comply with treatment and clinical management.
* Able to read and write English or Spanish.
* Consent of parent of guardian for patients under 18 years.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consenting patients newly enrolled in either CPCRA 007 or CPCRA 006
Sampling Method: Non-Probability Sample
Enrollment: 557 (Actual)
Dates: Start 1994-10; Primary Completion 1996-09 (Actual); Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Besch CL, Study Chair; Morse EV, Study Chair; Simon PM, Study Chair
Locations (13):
- United States (13):
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Simon PM, Morse EV, Besch L. Barriers to compliance among women co-enrolled in a PCP prophylaxis and compliance protocol. HIV Infect Women Conf. 1995 Feb 22-24:P109